CLINICAL TRIAL: NCT01688778
Title: The Copenhagen Rehabilitation Trial Part 2: Telemedicine as a Means to Achieve Good Diabetes Control Among Patients With Type 2 Diabetes
Brief Title: Telemedicine as a Means to Achieving Good Diabetes Control Among Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: The Health and Care Committee, Copenhagen City Council (Unknown)
Responsible Party: Principal Investigator, Caroline Raun Hansen, MD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-2-2011-158
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Type 2 Diabetes; Poor Glycemic Control; Medication Adherence
Keywords: Type 2 diabetes; Quality of life; Lifestyle intervention; Telemedicine; Videoconference
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine (Experimental): Monthly video consultations with a nurse as add-on to standard treatment.
  Interventions: Behavioral: Telemedicine
- Standard treatment (No Intervention): Standard diabetes control at a Diabetes Clinic or GP

INTERVENTIONS:
Behavioral: Telemedicine — Monthly video consultations with a nurse as add-on to standard treatment. The nurse has access to bloodsugar- bloodpressure and weight measurements uploaded by the participants to a tablet computer directly from the devices.
  Patients on Insulin measure bloodsugar twice a day (fasting and before their evening meal). Patients not on Insulin measure bloodsugar once a week (fasting and before their evening meal). All participants measure bloodpressure and weight once a week. The intervention lasts 32 weeks.
  Arms: Telemedicine

SUMMARY:
The aim of the study is to investigate the effect of telemedicine among the group of type-2-diabetics who, despite rehabilitation, remain poorly regulated. To describe the patients with regards to vulnerability and social resources and to determine wich groups benefit the most from telemedicine.

DETAILED DESCRIPTION:
Type-2-diabetes is a growing healthcare problem. Both because of the increasing amount of patients and because of the complications of diabetes.

Non-pharmacological treatment is considered fundamental in the treatment of patients with type-2-diabetes.

In the Community of Copenhagen, all patients diagnosed with diabetes receive rehabilitation. The rehabilitation consists of counseling with regards to nutrition, physical activity, smoking cessation and education about diabetes.

Some patients however, remain poorly regulated despite rehabilitation as well as pharmacological treatment.

A total number of 165 patients will be randomized to intervention group or standard care.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c > 7,5%
* BMI > 25
* Spoken danish
* Completed a rehabilitation program more than 6 months ago

Exclusion Criteria:

* HbA1c < 7,5%
* BMI < 25
* Need of interpreter

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-04-28 (Actual); Study Completion 2015-04-28 (Actual)

PRIMARY OUTCOMES:
Changes in HbA1c | Baseline, 16 weeks, 32 weeks, 6 months after intervention

SECONDARY OUTCOMES:
Fasting total cholesterol, LDL, HDL, triglycerides | Baseline, 32 weeks
Beta-cell function test (HOMA) | Baseline, 32 weeks
Weight | Baseline, 32 weeks
Bloodpressure | Baseline, 32 weeks
Physical activity | Baseline, 32 weeks
Change in quality of life | Baseline, 32 weeks
Waist circumference | Baseline, 32 weeks
Hip circumference | Baseline, 32 weeks
Body mass index | Baseline, 32 weeks
Use of medication | Baseline, 32 weeks

OTHER OUTCOMES:
Number of hospital admissions | 32 weeks
Number of visits at the emergency | 32 weeks
Number of visits at the outpatient department | 32 weeks
Number of visits at GP | 32-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Raun Hansen, MD, Principal Investigator — Endocrine Section, Bispebjerg Hospital, Bispebjerg Bakke 23, 2400 Copenhagen NV, Denmark
Locations (1):
- Endocrine Section, Dept. of Internal Medicine I, Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansen CR, Perrild H, Koefoed BG, Zander M. Video consultations as add-on to standard care among patients with type 2 diabetes not responding to standard regimens: a randomized controlled trial. Eur J Endocrinol. 2017 Jun;176(6):727-736. doi: 10.1530/EJE-16-0811. Epub 2017 Mar 21. PMID 28325823
- [Derived] Hansen CR, Perrild H, Koefoed BG, Faurschou P, Host D, Zander M. Effects of telemedicine in the treatment of patients with type 2 diabetes--a study protocol. Dan Med J. 2013 Dec;60(12):A4743. PMID 24355450